CLINICAL TRIAL: NCT01023581
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled Study to Determine the Efficacy and Safety of Alogliptin Plus Metformin, Alogliptin Alone, or Metformin Alone in Subjects With Type 2 Diabetes
Brief Title: Efficacy and Safety of Alogliptin Plus Metformin in Patients With Type 2 Diabetes
Acronym: AM7D
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SYR-322MET_302; 2009-012652-24 (Registry Identifier: EudraCT); U1111-1112-1912 (Registry Identifier: WHO); DOH-27-0910-3155 (Registry Identifier: SANCTR); CTRI/2010/091/000253 (Registry Identifier: CTRI)
Record Dates: First submitted 2009-12-01; First posted 2009-12-02 (Estimated); Results first posted 2013-03-26 (Estimated); Last update posted 2013-03-26 (Estimated); Status verified 2013-02

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Type 2 Diabetes mellitus; Non-insulin dependent diabetes mellitus; Drug Therapy; Hypoglycemia,; Hyperglycemia
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Hypoglycemia; Hyperglycemia | interventions — alogliptin; Metformin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (7):
- Placebo (Placebo Comparator): Alogliptin placebo-matching tablets, orally, twice daily and Metformin placebo-matching capsules, orally, twice daily for up to 26 weeks.
  Interventions: Drug: Alogliptin Placebo; Drug: Metformin Placebo
- Alogliptin 25 QD (Experimental): Alogliptin 25 mg, tablets, orally, once daily (QD) and Metformin placebo-matching capsules, orally, twice daily for up to 26 weeks.
  Interventions: Drug: Alogliptin; Drug: Metformin Placebo
- Alogliptin 12.5 BID (Experimental): Alogliptin 12.5 mg, tablets, orally, twice daily (BID) and Metformin placebo-matching capsules, orally, twice daily for up to 26 weeks.
  Interventions: Drug: Alogliptin; Drug: Metformin Placebo
- Metformin 500 BID (Active Comparator): Alogliptin placebo-matching tablets, orally, twice daily and Metformin 500 mg capsules, orally, twice daily for up to 26 weeks.
  Interventions: Drug: Metformin; Drug: Alogliptin Placebo
- Metformin 1000 BID (Active Comparator): Alogliptin placebo-matching tablets, orally, twice daily and Metformin 1000 mg capsules, orally, twice daily for up to 26 weeks.
  Interventions: Drug: Metformin; Drug: Alogliptin Placebo
- Alogliptin 12.5 BID + Metformin 500 BID (Experimental): Alogliptin 12.5mg, tablets, orally, twice daily and Metformin 500 mg, capsules, orally, twice daily for up to 26 weeks.
  Interventions: Drug: Alogliptin; Drug: Metformin
- Alogliptin 12.5 BID + Metformin 1000 BID (Experimental): Alogliptin 12.5 mg, tablets, orally, twice daily and Metformin 1000 mg, capsules, orally, twice daily for up to 26 weeks.
  Interventions: Drug: Alogliptin; Drug: Metformin

INTERVENTIONS:
Drug: Alogliptin — Alogliptin tablets.
  Other Names: SYR-322
  Arms: Alogliptin 12.5 BID; Alogliptin 12.5 BID + Metformin 1000 BID; Alogliptin 12.5 BID + Metformin 500 BID; Alogliptin 25 QD
Drug: Metformin — Metformin capsules
  Other Names: Glucophage; Glucophage XR; Riomet; Fortamet; Glumetza; Obimet; Dianben; Diabex; Diaformin
  Arms: Alogliptin 12.5 BID + Metformin 1000 BID; Alogliptin 12.5 BID + Metformin 500 BID; Metformin 1000 BID; Metformin 500 BID
Drug: Alogliptin Placebo — Alogliptin placebo-matching tablets.
  Arms: Metformin 1000 BID; Metformin 500 BID; Placebo
Drug: Metformin Placebo — Metformin placebo-matching capsules.
  Arms: Alogliptin 12.5 BID; Alogliptin 25 QD; Placebo

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of alogliptin combined with metformin, once daily (QD) or twice daily (BID), in participants with Type 2 Diabetes.

DETAILED DESCRIPTION:
There are approximately 19 million people in the United States who have been diagnosed with diabetes mellitus, of which 90% to 95% are type 2. The prevalence of type 2 diabetes varies among racial and ethnic populations and has been shown to correlate with age, obesity, family history, history of gestational diabetes and physical inactivity. Over the next decade, a marked increase in the number of adults with diabetes mellitus is expected.

Metformin is the usual choice of first-line therapy for type 2 diabetes. Metformin targets insulin resistance in type 2 diabetes by inhibiting hepatic glucose production and stimulating glucose uptake in skeletal muscle and adipose tissue, which results in a long-term glucose-lowering effect.

Alogliptin is an inhibitor of the dipeptidyl peptidase IV enzyme. Dipeptidyl peptidase-4 enzyme is thought to be primarily responsible for the in vivo degradation of 2 peptide hormones released in response to nutrient ingestion, namely glucagon-like peptide-1 and glucose-dependent insulinotropic peptide. Both peptides exert important effects on islet beta cells to stimulate glucose-dependent insulin secretion as well as regulating beta cell proliferation and cytoprotection. Glucagon-like peptide-1, but not glucose-dependent insulinotropic peptide, inhibits gastric emptying, glucagon secretion, and food intake. Glucose-dependent insulinotropic peptide has been shown to enhance insulin secretion by direct interaction with a glucose-dependent insulinotropic peptide -specific receptor on islet beta cells. The glucose-lowering actions of glucagon-like peptide-1, but not glucose-dependent insulinotropic peptide, are preserved in patients with type 2 diabetes mellitus. It is expected that inhibition of dipeptidyl peptidase IV will improve glycemic (glucose) control in patients with type 2 diabetes.

Based on the potential, complimentary mechanisms of action of alogliptin and metformin, this study will compare the safety and efficacy of alogliptin and metformin (SYR-322MET) on improving glycemic control in patients with type 2 diabetes mellitus who are inadequately controlled by diet adjustment and exercise alone.

Participants taking part in this study will receive dietary and exercise coaching, and will monitor their own blood glucose concentrations with a home glucose monitor. Participants will also be required to maintain a hypoglycemic diary throughout the course of the study. Participation in this study is expected to last up to 34 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Has historical diagnosis of Type 2 Diabetes Mellitus.
* Has been treated with diet and exercise for at least 2 months prior to Screening, and has a Glycosylated Hemoglobin concentration between 7.5% and 10.0%, inclusive at Screening.
* Has received less than 7 days of any antidiabetic medication within 2 months prior to Screening.
* Body mass index greater than or equal to 23 kg/m^2 and less than or equal to 45 kg/m^2 (except for Asian or Asian-descendant subjects for whom the range is between 20 and 35 kg/ m^2, inclusive).
* Fasting C-peptide concentration greater than or equal to 0.8 ng/mL.
* Regularly using other, non-excluded, medications must be on a stable dose for at least the 4 weeks prior to Screening.
* Females of childbearing potential and males who are sexually active agree to routinely use adequate contraception from Screening throughout the duration of the study.
* Able and willing to monitor their own blood glucose concentrations with a home glucose monitor and complete patient diaries.

Exclusion Criteria:

* Hemoglobin less than 12 g/dL for males and less than 10 g/dL for females at Screening Visit.
* Has a history of any hemoglobinopathy that may affect determination of Glycosylated Hemoglobin.
* Has a history of laser treatment for proliferative diabetic retinopathy within the 6 months prior to Screening.
* Has a history of treatment for diabetic gastric paresis, gastric banding, or gastric bypass surgery.
* Has a history of diabetic ketoacidosis or hyperosmolar non-ketotic coma.
* Has systolic blood pressure greater than or equal to 150 mmHg and /or diastolic pressure greater than or equal to 90 mmHg at Screening visit.
* Has New York Heart Association Class III to IV heart failure.
* Has a history of coronary angioplasty, coronary stent placement, coronary bypass surgery, or myocardial infarction within the 90 days prior to Screening.
* Has Alanine aminotransferase greater than 3 times the upper limit of normal at Screening.
* Has a history of alcohol or substance abuse with the 2 years prior to Screening.
* Serum creatinine greater than or equal to 1.5 mg/dL for males and greater than or equal to 1.4 mg/dL for females.
* Has history of cancer, other than squamous cell or basal cell carcinoma of the skin that has not been in full remission for at least 5 years prior to Screening.
* Has a history of infection with human immunodeficiency virus, hepatitis B virus or hepatitis C virus.
* Has any major illness or debility that in the investigator's opinion prohibits the subject from completing the study.
* Has received any investigational drug within the 90 days prior to Screening.
* Has a history of hypersensitivity or allergy to alogliptin, other DPP-4 inhibitors, metformin or related compounds.
* Has used oral or systematically injected glucocorticoids or weight loss drugs prior to 2 months to screening.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 784 (Actual)
Dates: Start 2009-11; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vice President, Clinical Science, Study Director — Takeda
Locations (201):
- United States (109):
  - Dothan, Alabama
  - Muscle Shoals, Alabama
  - Pell City, Alabama
  - Chandler, Arizona
  - Mesa, Arizona
  - Phoenix, Arizona
  - Sierra Vista, Arizona
  - Tempe, Arizona
  - Little Rock, Arkansas
  - Searcy, Arkansas
  - Tempe, Arkansas
  - Anaheim, California
  - Buena Park, California
  - Cathedral City, California
  - National City, California
  - Pismo Beach, California
  - Roseville, California
  - Santa Ana, California
  - Colorado Springs, Colorado
  - Boca Raton, Florida
  - Bradenton, Florida
  - Cutler Bay, Florida
  - Hialeah, Florida
  - Lauderdale Lakes, Florida
  - Miami, Florida
  - Ocala, Florida
  - Opa-locka, Florida
  - Orlando, Florida
  - Panama City, Florida
  - Pembroke Pines, Florida
  - Atlanta, Georgia
  - Blue Ridge, Georgia
  - Decatur, Georgia
  - Lawrenceville, Georgia
  - Hayden Lake, Idaho
  - Chicago, Illinois
  - Melrose Park, Illinois
  - La Porte, Indiana
  - Mishawaka, Indiana
  - Council Bluffs, Iowa
  - Dubuque, Iowa
  - Topeka, Kansas
  - Lexington, Kentucky
  - Louisville, Kentucky
  - Marrero, Louisiana
  - Oxon Hill, Maryland
  - North Dartmouth, Massachusetts
  - Dearborn, Michigan
  - Flint, Michigan
  - Kalamazoo, Michigan
  - Picayune, Mississippi
  - St Louis, Missouri
  - Omaha, Nebraska
  - Henderson, Nevada
  - Las Vegas, Nevada
  - Brick, New Jersey
  - Elizabeth, New Jersey
  - North Massapequa, New York
  - Asheville, North Carolina
  - Charlotte, North Carolina
  - Greensboro, North Carolina
  - Mooresville, North Carolina
  - Fargo, North Dakota
  - Cincinnati, Ohio
  - Cleveland, Ohio
  - Gallipolis, Ohio
  - Mason, Ohio
  - Maumee, Ohio
  - Norman, Oklahoma
  - Oklahoma City, Oklahoma
  - Tulsa, Oklahoma
  - Altoona, Pennsylvania
  - Bensalem, Pennsylvania
  - Downingtown, Pennsylvania
  - Fleetwood, Pennsylvania
  - Perkasie, Pennsylvania
  - Shippensburg, Pennsylvania
  - Tipton, Pennsylvania
  - Uniontown, Pennsylvania
  - Columbia, South Carolina
  - Greenville, South Carolina
  - Murrells Inlet, South Carolina
  - North Myrtle Beach, South Carolina
  - Taylors, South Carolina
  - Brentwood, Tennessee
  - Bristol, Tennessee
  - Crossville, Tennessee
  - Johnson City, Tennessee
  - McKenzie, Tennessee
  - Spring Hill, Tennessee
  - Carrollton, Texas
  - Dallas, Texas
  - Deer Park, Texas
  - El Paso, Texas
  - Houston, Texas
  - Hurst, Texas
  - Katy, Texas
  - Odessa, Texas
  - San Antonio, Texas
  - Schertz, Texas
  - Spring, Texas
  - Sugarland, Texas
  - Temple, Texas
  - Bountiful, Utah
  - Ogden, Utah
  - Salt Lake City, Utah
  - South Burlington, Vermont
  - Petersburg, Virginia
  - Milwaukee, Wisconsin
- Czechia (6):
  - Hradec Králové
  - Olomouc
  - Ostrava
  - Prague
  - Zlín
  - Znojmo
- Hungary (8):
  - Budaörs
  - Debrecen
  - Gyöngyös
  - Győr
  - Gyula
  - Komárom
  - Szolnok
  - Zalaegerszeg
- Israel (5):
  - Haifa
  - Holon
  - Kfar Saba
  - Nahariya
  - Safed
- Lithuania (4):
  - Kaunas
  - Kėdainiai
  - Klaipėda
  - Vilnius
- Mexico (17):
  - Acapulco, Guerrero
  - Cuernavaca
  - Culiacan, Sinoloa
  - Distrito Federal
  - Durango
  - Durango, Durango
  - Guadalajara
  - Mexico City
  - Mexico City, Mexico
  - Monclova, Coahuila
  - Monterrey
  - Monterrey, NL
  - Pachuca
  - Pachuca, Hidalgo
  - Saltillo
  - Tijuana, Baja California
  - Zapopan, Jalisco
- Poland (8):
  - Bialystok
  - Bytom
  - Gniewkowo
  - Grodzisk Mazowiecki
  - Kamieniec Ząbkowicki
  - Warsaw
  - Wroclaw
  - Łęczyca
- Puerto Rico (8):
  - Caguas, PR
  - Cidra, PR
  - Ponce, PR
  - Salinas, PR
  - San Juan, PR
  - Santurce, PR
  - San Juan
  - Trujilo Alto
- Romania (6):
  - Bacau
  - Baia Mare
  - Bucharest
  - Constanța
  - Iași
  - Ploieşti
- Russia (7):
  - Arkhangelsk
  - Irkutsk
  - Kemerovo
  - Moscow
  - Perm
  - Saint Petersburg
  - Ufa
- Slovakia (8):
  - Banská Bystrica
  - Košice
  - Lučenec
  - Nitra
  - Prešov
  - Prievidza
  - Šahy
  - Žilina
- South Africa (6):
  - Centurion, Gauteng
  - Johannesburg, Gauteng
  - Pretoria, Gauteng
  - Durban, KwaZulu-Natal
  - Cape Town, Western Cape
  - Pretoria
- Ukraine (9):
  - Dnipropetrovsk
  - Donetsk
  - Ivano-Frankivsk
  - Kharkiv
  - Kyiv
  - Lviv
  - Odesa
  - Vinnytsia
  - Zaporizhzhya

REFERENCES:
- [Derived] Pratley RE, Fleck P, Wilson C. Efficacy and safety of initial combination therapy with alogliptin plus metformin versus either as monotherapy in drug-naive patients with type 2 diabetes: a randomized, double-blind, 6-month study. Diabetes Obes Metab. 2014 Jul;16(7):613-21. doi: 10.1111/dom.12258. Epub 2014 Feb 12. PMID 24400655

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 198 investigative sites worldwide from 16 November 2009 to 30 June 2011.
Pre-assignment Details: Participants with a diagnosis of type 2 diabetes and glycemia inadequately controlled on diet and exercise alone were randomly assigned with equal probability to 1 of 7 treatment groups, including placebo, alogliptin alone, metformin alone or a combination of alogliptin and metformin.
Period: Overall Study
Arm/Group | Placebo | Alogliptin 25 QD | Alogliptin 12.5 BID | Metformin 500 BID | Metformin 1000 BID | Alogliptin 12.5 BID + Metformin 500 BID | Alogliptin 12.5 BID + Metformin 1000 BID
Started | 109 | 112 | 113 | 114 | 111 | 111 | 114
Received Study Treatment | 106 | 112 | 110 | 109 | 111 | 106 | 114
Completed | 74 (The number of completed patients represents those who completed study drug.) | 89 | 71 | 94 | 95 | 92 | 94
Not Completed | 35 | 23 | 42 | 20 | 16 | 19 | 20
Not completed — Adverse Event | 4 | 4 | 7 | 3 | 2 | 5 | 11
Not completed — Major protocol deviation | 2 | 0 | 3 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 4 | 8 | 7 | 2 | 5 | 2 | 2
Not completed — Withdrawal by Subject | 13 | 8 | 16 | 10 | 6 | 8 | 5
Not completed — Pregnancy | 0 | 0 | 0 | 2 | 0 | 1 | 0
Not completed — Lack of Efficacy | 9 | 3 | 6 | 2 | 1 | 2 | 1
Not completed — Physician Decision | 2 | 0 | 2 | 1 | 1 | 1 | 1
Not completed — Other | 1 | 0 | 1 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Alogliptin 25 QD | Alogliptin 12.5 BID | Metformin 500 BID | Metformin 1000 BID | Alogliptin 12.5 BID + Metformin 500 BID | Alogliptin 12.5 BID + Metformin 1000 BID | Total
Number analyzed (Participants) | 109 | 112 | 113 | 114 | 111 | 111 | 114 | 784
Age Continuous [Mean (Standard Deviation); unit: years] | 53.1 (9.60) | 52.6 (9.38) | 53.7 (9.70) | 54.6 (10.20) | 52.6 (11.30) | 53.7 (11.59) | 54.6 (10.42) | 53.5 (10.33)
Age, Customized [Number; unit: participants]
  <65 years | 100 | 103 | 96 | 95 | 94 | 91 | 96 | 675
  ≥65 years | 9 | 9 | 17 | 19 | 17 | 20 | 18 | 109
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 54 | 64 | 50 | 67 | 60 | 63 | 52 | 410
  Male | 55 | 48 | 63 | 47 | 51 | 48 | 62 | 374
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic or Latino | 45 | 43 | 43 | 45 | 42 | 45 | 39 | 302
  Not Hispanic or Latino | 64 | 69 | 70 | 69 | 69 | 66 | 75 | 482
Race/Ethnicity, Customized [Number; unit: participants]
  American Indian or Alaska Native | 5 | 8 | 5 | 3 | 6 | 9 | 5 | 41
  Asian | 20 | 17 | 21 | 19 | 20 | 20 | 26 | 143
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
  Black or African American | 8 | 3 | 3 | 6 | 6 | 6 | 5 | 37
  White | 76 | 84 | 83 | 85 | 79 | 76 | 78 | 561
  Multiracial | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 31.15 (5.269) | 30.81 (5.219) | 30.36 (5.159) | 30.19 (4.842) | 30.51 (5.043) | 30.92 (5.353) | 31.04 (5.375) | 30.71 (5.173)
Diabetes Duration [Mean (Standard Deviation); unit: years] | 4.25 (4.778) | 3.65 (4.119) | 3.97 (4.800) | 3.78 (3.904) | 4.08 (4.587) | 4.13 (4.777) | 4.22 (4.972) | 4.01 (4.563)
Baseline HbA1c [Number; unit: participants] — The count for baseline HbA1c category is based on HbA1c value used in randomization for stratification.
  participants
    ≤8.5% | 65 | 67 | 67 | 67 | 66 | 66 | 67 | 465
    >8.5% | 44 | 45 | 46 | 47 | 45 | 45 | 47 | 319

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Glycosylated Hemoglobin (HbA1c) at Week 26
Description: The change from Baseline to Week 26 in HbA1c (the concentration of glucose bound to hemoglobin as a percent of the absolute maximum that can be bound).
Time Frame: Baseline and Week 26.
Population: Full analysis set (patients who took at least 1 dose of study medication) where baseline and at least 1 postbaseline assessment were available. Analysis includes only data collected on or after baseline and within 7 days after last dose of study medication or hyperglycemic rescue, whichever came first. Last observation carried forward was utilized.
Measure: Least Squares Mean (Standard Error); unit: percentage glycosylated hemoglobin
Arm/Group | Placebo | Alogliptin 25 QD | Alogliptin 12.5 BID | Metformin 500 BID | Metformin 1000 BID | Alogliptin 12.5 BID + Metformin 500 BID | Alogliptin 12.5 BID + Metformin 1000 BID
Number analyzed (Participants) | 102 | 104 | 104 | 103 | 108 | 102 | 111
percentage glycosylated hemoglobin | 0.15 (0.094) | -0.52 (0.094) | -0.56 (0.093) | -0.65 (0.094) | -1.11 (0.092) | -1.22 (0.094) | -1.55 (0.090)
Statistical Analysis 1: Comparison: Alogliptin 12.5 BID vs Alogliptin 12.5 BID + Metformin 500 BID; The primary efficacy analysis consisted of 2 separate sets of comparisons between each BID combination of alogliptin and metformin (alogliptin/metformin 12.5/500 mg BID and 12.5/1000 mg BID) and its constituent doses of alogliptin and metformin. The null hypothesis was that the combination of alogliptin and metformin had no additional effect on glycemic control at Week 26 either when compared with the constituent dose of alogliptin or with the constituent dose of metformin; Test type: Superiority or Other; p < 0.001, ANCOVA — For each set of comparisons in the primary analysis, the null hypothesis was rejected only if both comparisons between a combination and its constituent doses were statistically significant at the 2-sided 2.5% level; ANCOVA model with treatment and geographic region as fixed effects and baseline HbA1c as a covariate; LS mean difference = -0.67, 95% CI 2-sided [-0.96 to -0.37]
Statistical Analysis 2: Comparison: Metformin 500 BID vs Alogliptin 12.5 BID + Metformin 500 BID; Test type: Superiority or Other; p < 0.001, ANCOVA; ANCOVA model with treatment and geographic region as fixed effects and baseline HbA1c as a covariate; LS mean difference = -0.57, 95% CI 2-sided [-0.87 to -0.27]
Statistical Analysis 3: Comparison: Alogliptin 12.5 BID vs Alogliptin 12.5 BID + Metformin 1000 BID; Test type: Superiority or Other; p < 0.001, ANCOVA; ANCOVA model with treatment and geographic region as fixed effects and baseline HbA1c as a covariate; LS mean difference = -1.00, 95% CI 2-sided [-1.29 to -0.71]
Statistical Analysis 4: Comparison: Metformin 1000 BID vs Alogliptin 12.5 BID + Metformin 1000 BID; Test type: Superiority or Other; p < 0.001, ANCOVA; ANCOVA model with treatment and geographic region as fixed effects and baseline HbA1c as a covariate; LS mean difference = -0.44, 95% CI 2-sided [-0.73 to -0.16]

2. Secondary Outcome: Change From Baseline in HbA1c Over Time
Description: The change from Baseline in HbA1c (the concentration of glucose bound to hemoglobin as a percent of the absolute maximum that can be bound) was assessed at Weeks 4, 8, 12, 16 and 20.
  Least squares means are from an analysis of covariance (ANCOVA) model with treatment and geographic region as fixed effects, and baseline HbA1c as a covariate.
Time Frame: Baseline and Weeks 4, 8, 12, 16, and 20.
Population: The full analysis set where a baseline assessment and at least 1 valid postbaseline assessment were available. The analysis includes only data collected on or after baseline and within 7 days after the last dose of study medication or hyperglycemic rescue, whichever came first. Last observation carried forward was utilized.
Measure: Least Squares Mean (Standard Error); unit: percentage glycosylated hemoglobin
Arm/Group | Placebo | Alogliptin 25 QD | Alogliptin 12.5 BID | Metformin 500 BID | Metformin 1000 BID | Alogliptin 12.5 BID + Metformin 500 BID | Alogliptin 12.5 BID + Metformin 1000 BID
Number analyzed (Participants) | 106 | 112 | 110 | 109 | 111 | 106 | 114
percentage glycosylated hemoglobin
  Week 4 (n=95, 97, 89, 94, 102, 94, 101) | 0.09 (0.058) | -0.34 (0.057) | -0.42 (0.060) | -0.37 (0.058) | -0.58 (0.056) | -0.70 (0.058) | -0.75 (0.056)
  Week 8 (n=102, 104, 104, 103, 108, 102, 111) | 0.08 (0.073) | -0.51 (0.073) | -0.58 (0.072) | -0.59 (0.073) | -0.86 (0.071) | -1.08 (0.073) | -1.17 (0.070)
  Week 12 (n=102, 104, 104, 103, 108, 102, 111) | 0.12 (0.081) | -0.53 (0.080) | -0.62 (0.080) | -0.68 (0.081) | -1.02 (0.079) | -1.22 (0.081) | -1.40 (0.078)
  Week 16 (n=102, 104, 104, 103, 108, 102, 111) | 0.13 (0.087) | -0.58 (0.087) | -0.63 (0.086) | -0.72 (0.087) | -1.09 (0.085) | -1.26 (0.087) | -1.50 (0.084)
  Week 20 (n=102, 104, 104, 103, 108, 102, 111) | 0.12 (0.092) | -0.57 (0.091) | -0.59 (0.091) | -0.68 (0.092) | -1.14 (0.089) | -1.25 (0.092) | -1.54 (0.088)

3. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose Over Time
Description: The change from Baseline in fasting plasma glucose was assessed at Weeks 1, 2, 4, 8, 12, 16, 20 and 26. Least Squares Means were from an ANCOVA model with treatment and geographic region as fixed effects, and baseline fasting plasma glucose as a covariate.
Time Frame: Baseline and Weeks 1, 2, 4, 8, 12, 16, 20 and 26.
Population: Full analysis set where a baseline assessment and at least 1 valid postbaseline assessment were available. Includes only data collected on or after baseline and within 1 day after the last dose of study medication or hyperglycemic rescue, whichever came first. Last observation carried forward was utilized.
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Placebo | Alogliptin 25 QD | Alogliptin 12.5 BID | Metformin 500 BID | Metformin 1000 BID | Alogliptin 12.5 BID + Metformin 500 BID | Alogliptin 12.5 BID + Metformin 1000 BID
Number analyzed (Participants) | 106 | 112 | 110 | 109 | 111 | 106 | 114
mg/dL
  Week 1 (n=102, 103, 94, 95, 104, 101, 109) | 5.7 (3.40) | -3.9 (3.38) | -11.9 (3.54) | -12.6 (3.52) | -23.1 (3.36) | -32.7 (3.41) | -36.3 (3.29)
  Week 2 (n=105, 112, 105, 102, 108, 106, 111) | 4.6 (3.58) | -7.4 (3.46) | -11.6 (3.58) | -14.5 (3.63) | -22.2 (3.53) | -34.5 (3.56) | -43.6 (3.48)
  Week 4 (n=105, 112, 106, 106, 110, 106, 111) | 7.2 (3.69) | -11.5 (3.57) | -16.6 (3.67) | -16.9 (3.67) | -29.0 (3.60) | -37.6 (3.67) | -44.1 (3.58)
  Week 8 (n=105, 112, 106, 106, 110, 106, 112) | 7.1 (4.00) | -10.9 (3.87) | -12.1 (3.98) | -11.8 (3.98) | -30.7 (3.91) | -32.9 (3.98) | -43.8 (3.87)
  Week 12 (n=105, 112, 106, 106, 110, 106, 112) | 11.6 (4.16) | -9.7 (4.03) | -14.7 (4.14) | -14.0 (4.14) | -30.7 (4.06) | -31.6 (4.14) | -44.7 (4.03)
  Week 16 (n=105, 112, 106, 106, 110, 106, 112) | 10.1 (4.17) | -7.1 (4.04) | -14.7 (4.15) | -13.3 (4.15) | -33.5 (4.07) | -35.9 (4.15) | -47.7 (4.04)
  Week 20 (n=105, 112, 106, 106, 110, 106, 112) | 8.7 (4.36) | -9.2 (4.22) | -12.3 (4.34) | -10.9 (4.34) | -35.1 (4.25) | -33.8 (4.34) | -44.6 (4.22)
  Week 26 (n=105, 112, 106, 106, 110, 106, 112) | 12.4 (4.52) | -6.1 (4.37) | -9.7 (4.49) | -11.5 (4.49) | -31.9 (4.41) | -31.7 (4.49) | -45.9 (4.37)

ADVERSE EVENTS:
Time Frame: Adverse events that occurred after the first dose of double-blind study medication and within 14 days after the last dose of double-blind study medication.
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Placebo | Alogliptin 25 QD | Alogliptin 12.5 BID | Metformin 500 BID | Metformin 1000 BID | Alogliptin 12.5 BID + Metformin 500 BID | Alogliptin 12.5 BID + Metformin 1000 BID
Serious Adverse Events (participants affected / at risk) | 3/106 | 1/112 | 4/110 | 3/109 | 2/111 | 2/106 | 2/114
Other Adverse Events (participants affected / at risk) | 50/106 | 38/112 | 34/110 | 44/109 | 43/111 | 40/106 | 37/114
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=106) | Alogliptin 25 QD (N=112) | Alogliptin 12.5 BID (N=110) | Metformin 500 BID (N=109) | Metformin 1000 BID (N=111) | Alogliptin 12.5 BID + Metformin 500 BID (N=106) | Alogliptin 12.5 BID + Metformin 1000 BID (N=114)
Angina pectoris (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Myocardial ischaemia (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Wandering pacemaker (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Gallbladder empyema (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Ischaemic stroke (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Tremor (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Multiple drug overdose intentional (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Alveolitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Delusion (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Urinary retention (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=106) | Alogliptin 25 QD (N=112) | Alogliptin 12.5 BID (N=110) | Metformin 500 BID (N=109) | Metformin 1000 BID (N=111) | Alogliptin 12.5 BID + Metformin 500 BID (N=106) | Alogliptin 12.5 BID + Metformin 1000 BID (N=114)
Hyperglycaemia (Metabolism and nutrition disorders) | 28 | 19 | 13 | 19 | 9 | 8 | 1
Headache (Nervous system disorders) | 3 | 6 | 5 | 8 | 4 | 7 | 6
Diarrhoea (Gastrointestinal disorders) | 3 | 1 | 3 | 4 | 10 | 6 | 8
Dyslipidaemia (Metabolism and nutrition disorders) | 6 | 1 | 2 | 7 | 6 | 6 | 2
Hypertension (Vascular disorders) | 5 | 3 | 2 | 6 | 1 | 5 | 8
Creatinine renal clearance decreased (Investigations) | 4 | 1 | 4 | 0 | 6 | 5 | 9
Upper respiratory tract infection (Infections and infestations) | 3 | 3 | 3 | 4 | 3 | 8 | 2
Nausea (Gastrointestinal disorders) | 2 | 0 | 3 | 4 | 6 | 3 | 6
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 3 | 3 | 1 | 3 | 6 | 6 | 1
Nasopharyngitis (Infections and infestations) | 2 | 7 | 1 | 2 | 4 | 3 | 2
Dyspepsia (Gastrointestinal disorders) | 3 | 0 | 1 | 0 | 2 | 0 | 8
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 6 | 1 | 4 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.